CLINICAL TRIAL: NCT04252443
Title: Nurses' Knowledge and Attitudes Towards Opioids in Pain Management in North Cyprus
Brief Title: Nurses' Knowledge and Attitude About Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Principal Investigator, Semra Aslay, Ass. Prof. (M.D.), European University of Lefke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: opioid
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Opioid Use, Unspecified; Nurse's Role; Knowledge, Attitudes, Practice
Keywords: Opioid; Knowledge; Attitude; Nursing
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: The research population consisted of 190 nurses working in a university hospital. Because all of the nurses in the research population could not be reached, a sample was selected using a simple random sampling method. One hundred twenty-seven nurses were interviewed in the research population, with a 95% confidence interval and a 5% sampling error.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurse (Other): The research population consisted of 190 nurses working in a university hospital. Because all of the nurses in the research population could not be reached, a sample was selected using a simple random sampling method. One hundred twenty-seven nurses were interviewed in the research population, with a 95% confidence interval and a 5% sampling error.
  Interventions: Other: Evaluation of nurses' knowledge and attitudes about opioid analgesics working in a university hospital

INTERVENTIONS:
Other: Evaluation of nurses' knowledge and attitudes about opioid analgesics working in a university hospital — Interventions involving nurses' pharmacological level
  Other Names: Knowledge about opioid and adjuvant analgesics; Opinions and attitudes on opioid administration

SUMMARY:
Opioid analgesics used in moderate or severe pain have potential side effects and addiction. Therefore, nurses have hesitations about opioid administration.This descriptive study aimed to evaluate the attitude and knowledge of nurses working in a university hospital about opioids. One hundred twenty-seven nurses were interviewed in the research population. The research data were obtained from the questionnaire, prepared by the researchers, between 01-05 June 2018. It consisted of three parts: descriptive characteristics, attitudes, and knowledge on opioid administration, and evaluation of basic nursing skills and pharmacology about opioids. Statistical Package for Social Sciences (SPSS) 24.0 package program was used for statistical analysis.

DETAILED DESCRIPTION:
Analgesics do not eliminate the cause of pain but reduce or eliminate that feeling. Non-steroid analgesics are preferred in mild and moderate, and opioids are used to moderate or severe pain that does not respond to anti-inflammatory agents. However, nurses avoid the administration of opioids because of side effects and addiction risk.The first step in the effectiveness of pain management in the emergency department is evaluation and control. Pain control should be included in the emergency management system from the stage of triage assessment of the patient and should be concluded with the correct analgesic use, if necessary. In emergency departments, waiting for analgesia can be prolonged unnecessarily, and mostly insufficient doses of analgesics administered.Mainly the use of opioids in the emergency department is not preferred much because it reduces the symptoms and masks the examination findings. However, against this conventional idea, recent studies have shown that opioids use reduces pain-related anxiety.Also, it increases the patients' participation in the examination, thus making it more effective. While patients feel better, symptoms such as tenderness and defense were generally not affected by analgesia.This descriptive study was conducted to evaluate the attitude and knowledge of nurses working in a university hospital about opioid analgesic administration, after the ethical committee approved.

ELIGIBILITY:
Inclusion Criteria: Nurses, working university hospital, accepted to join to study

-

Exclusion Criteria:

* Other health care personnel, did not accept to join to study, long term leaving from job

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Nurses' Knowledge and Attitudes towards Opioids in Pain Management in North Cyprus | Through study completion, an average of 6 months
  Questionnaire, Knowledge scores of the participants were calculated over 100. 4 points were given for each correct answer, and 0 for each wrong or "don't know. " The range of scores was 0-100. A high score was a mean high level of knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Aslay, MD, Study Director — European University of Lefke
Locations (1):
- European University of Lefke, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participating data
Supporting Information: SAP
Time Frame: After published there is no ending frame
Access Criteria: Nurses working in university hospital in Northern Cyprus included in the study. In the research, a sample was selected using a simple random sampling method. One hundred twenty-seven nurses were interviewed in the research population, with a 95% confidence interval and a 5% sampling error.

REFERENCES:
- [Background] Abdolrazaghnejad A, Banaie M, Tavakoli N, Safdari M, Rajabpour-Sanati A. Pain Management in the Emergency Department: a Review Article on Options and Methods. Adv J Emerg Med. 2018 Jun 24;2(4):e45. doi: 10.22114/AJEM.v0i0.93. eCollection 2018 Fall. PMID 31172108
- [Background] Reagan KML, O'Sullivan DM, Gannon R, Steinberg AC. Decreasing postoperative narcotics in reconstructive pelvic surgery: a randomized controlled trial. Am J Obstet Gynecol. 2017 Sep;217(3):325.e1-325.e10. doi: 10.1016/j.ajog.2017.05.041. Epub 2017 May 25. PMID 28551445
- [Background] Janati M, Kariman H, Memary E, Davarinezhad-Moghadam E, Arhami-Dolatabadi A. Educational Intervention Effect on Pain Management Quality in Emergency Department; a Clinical Audit. Adv J Emerg Med. 2018 Jan 16;2(2):e16. doi: 10.22114/AJEM.v0i0.45. eCollection 2018 Spring. PMID 31172079
- [Background] Fein JA, Zempsky WT, Cravero JP; Committee on Pediatric Emergency Medicine and Section on Anesthesiology and Pain Medicine; American Academy of Pediatrics. Relief of pain and anxiety in pediatric patients in emergency medical systems. Pediatrics. 2012 Nov;130(5):e1391-405. doi: 10.1542/peds.2012-2536. Epub 2012 Oct 29. PMID 23109683
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Costello M, Thompson S. Preventing Opioid Misuse and Potential Abuse: The Nurse's Role in Patient Education. Pain Manag Nurs. 2015 Aug;16(4):515-9. doi: 10.1016/j.pmn.2014.09.008. Epub 2014 Dec 8. PMID 25497402
- [Background] Hunold KM, Esserman DA, Isaacs CG, Dickey RM, Pereira GF, Fillingim RB, Sloane PD, McLean SA, Platts-Mills TF. Side effects from oral opioids in older adults during the first week of treatment for acute musculoskeletal pain. Acad Emerg Med. 2013 Sep;20(9):872-9. doi: 10.1111/acem.12212. Epub 2013 Aug 27. PMID 24033733
- [Background] Trescot AM, Helm S, Hansen H, Benyamin R, Glaser SE, Adlaka R, Patel S, Manchikanti L. Opioids in the management of chronic non-cancer pain: an update of American Society of the Interventional Pain Physicians' (ASIPP) Guidelines. Pain Physician. 2008 Mar;11(2 Suppl):S5-S62. PMID 18443640
- [Background] Chapman CR, Lipschitz DL, Angst MS, Chou R, Denisco RC, Donaldson GW, Fine PG, Foley KM, Gallagher RM, Gilson AM, Haddox JD, Horn SD, Inturrisi CE, Jick SS, Lipman AG, Loeser JD, Noble M, Porter L, Rowbotham MC, Schoelles KM, Turk DC, Volinn E, Von Korff MR, Webster LR, Weisner CM. Opioid pharmacotherapy for chronic non-cancer pain in the United States: a research guideline for developing an evidence-base. J Pain. 2010 Sep;11(9):807-29. doi: 10.1016/j.jpain.2010.02.019. Epub 2010 Apr 28. PMID 20430701
- [Background] Gomes T, Tadrous M, Mamdani MM, Paterson JM, Juurlink DN. The Burden of Opioid-Related Mortality in the United States. JAMA Netw Open. 2018 Jun 1;1(2):e180217. doi: 10.1001/jamanetworkopen.2018.0217. PMID 30646062
- [Background] Hsaio GY, Chen IJ, Yu S, Wei IL, Fang YY, Tang FI. Nurses' knowledge of high-alert medications: instrument development and validation. J Adv Nurs. 2010 Jan;66(1):177-90. doi: 10.1111/j.1365-2648.2009.05164.x. PMID 20423443
- [Background] Samarkandi OA. Knowledge and attitudes of nurses toward pain management. Saudi J Anaesth. 2018 Apr-Jun;12(2):220-226. doi: 10.4103/sja.SJA_587_17. PMID 29628831
- [Background] de Freitas GR, de Castro CG Jr, Castro SM, Heineck I. Degree of knowledge of health care professionals about pain management and use of opioids in pediatrics. Pain Med. 2014 May;15(5):807-19. doi: 10.1111/pme.12332. Epub 2014 Jan 8. PMID 24401078
- [Background] Gorawara-Bhat R, Wong A, Dale W, Hogan T. Nurses' perceptions of pain management for older-patients in the Emergency Department: A qualitative study. Patient Educ Couns. 2017 Feb;100(2):231-241. doi: 10.1016/j.pec.2016.08.019. Epub 2016 Aug 29. PMID 27591825
- [Background] Charalambous A, Zorpas M, Cloconi C, Kading Y. Healthcare professionals' perceptions on the use of opioid analgesics for the treatment of cancer-related pain in Cyprus: A mixed-method study. SAGE Open Med. 2019 Apr 4;7:2050312119841823. doi: 10.1177/2050312119841823. eCollection 2019. PMID 31057793
- [Background] Tomaszek L, Debska G. Knowledge, compliance with good clinical practices and barriers to effective control of postoperative pain among nurses from hospitals with and without a "Hospital without Pain" certificate. J Clin Nurs. 2018 Apr;27(7-8):1641-1652. doi: 10.1111/jocn.14215. Epub 2018 Mar 2. PMID 29218814
- [Background] Al-Shaer D, Hill PD, Anderson MA. Nurses' knowledge and attitudes regarding pain assessment and intervention. Medsurg Nurs. 2011 Jan-Feb;20(1):7-11. PMID 21446289
- [Background] Hroch J, VanDenKerkhof EG, Sawhney M, Sears N, Gedcke-Kerr L. Knowledge and Attitudes about Pain Management among Canadian Nursing Students. Pain Manag Nurs. 2019 Aug;20(4):382-389. doi: 10.1016/j.pmn.2018.12.005. Epub 2019 May 15. PMID 31103502
- [Background] Peker L, Celebi N, Canbay O, Sahin A, Cakir B, Uzun S, Aypar U. Doctors' opinions, knowledge and attitudes towards cancer pain management in a university hospital. Agri. 2008 Apr;20(2):20-30. PMID 19021007
- [Background] Textor LH, Porock D. The pain management knowledge of nurses practicing in a rural midwest retirement community. J Nurses Staff Dev. 2006 Nov-Dec;22(6):307-12. doi: 10.1097/00124645-200611000-00007. PMID 17149048
- [Background] Kastanias P, Snaith KE, Robinson S. Patient-controlled oral analgesia: a low-tech solution in a high-tech world. Pain Manag Nurs. 2006 Sep;7(3):126-32. doi: 10.1016/j.pmn.2006.06.003. PMID 16931418
- [Background] Akbas M, Oztunc G. Examination of knowledge about and nursing interventions for the care of patients in pain of nurses who work at Cukurova University medical faculty Balcali hospital. Pain Manag Nurs. 2008 Sep;9(3):88-95. doi: 10.1016/j.pmn.2008.02.004. PMID 18706379
- [Background] Karaman E, Vural Dogru B, Yildirim Y. Knowledge and attitudes of nursing students about pain management. Agri. 2019 Apr;31(2):70-78. doi: 10.5505/agri.2018.10437. PMID 30995323
- See also: World Health Organization Analgesic Ladder Scheme — http://www.who.int/cancer/palliative/painladder/en/